CLINICAL TRIAL: NCT06909097
Title: MOV'D Strength Snacks vs Walk Breaks Study: Health Performance Gains Across Domains
Brief Title: Better Breaks: Strength Breaks vs Walk Breaks for Sedentary Behavior Breaks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marily Ann Oppezzo, Instructor Medicine - Med/Stanford Prevention Research Center, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 73022
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-09

CONDITIONS: Sedentary Employees
Keywords: physical activity breaks; prolonged sitting breaks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strength Snacks (Experimental): Participants will do 4 strength snacks throughout each work day, 2 of them post-prandial if possible.
  Interventions: Behavioral: Sitting breaks
- Walk Snacks (Active Comparator): Participants will take 4 x2 minute walk breaks throughout the sedentary workday, two of them post-prandial if possible.
  Interventions: Behavioral: Sitting breaks

INTERVENTIONS:
Behavioral: Sitting breaks — Participants will take 2 minute physical movement breaks throughout a sedentary work day.

SUMMARY:
This study investigates the benefits of two different types of 2 minute activity breaks during sedentary workdays for people who sit for long periods of time in sedentary jobs.

DETAILED DESCRIPTION:
For this study, participants are randomly assigned to one of two physical activity breaks and for 8 weeks are to do 4 per day and track their daily breaks and productivity. There are many measurements including: in-person strength assessments at baseline, 1 month, and 2 months; daily tracking of breaks; pre and post oral glucose tolerance tests; pre and post 10-day diet tracking; pre and post 10-day Continuous Glucose Monitoring with a Dexcom; genome with saliva at pre; and -omics at pre and post.

ELIGIBILITY:
Inclusion Criteria:

-

Identify inclusion criteria.

1. Sedentary occupation (e.g., clerical work, data entry, call center, receptionists)
2. Full time employment remote or on-site
3. Able to safely perform bodyweight squats and lunges
4. Over 30 years old
5. Not currently doing a strength training program
6. Not currently taking planned activity breaks at work
7. Has a smart phone with a camera and unlimited text plans
8. Interested in participating
9. Fluent in English
10. Not currently on insulin or any glucose lowering medication

Exclusion Criteria:

1. Yes to any of the physical activity readiness criteria questionnaire (e.g. cardiac symptoms with increasing heart rate, dizziness upon performing exercise)
2. Participating in another research study on diet, weight loss, or any physical activity.
3. If their doctor has ever said to not strength train
4. Having insulin dependence

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in average area under the curve for glucose from a 10 day continuous glucose monitors | from baseline to post (8 weeks)
  Change from pre to post in average area under the curve for glucose from a 10 day continuous glucose monitors

SECONDARY OUTCOMES:
Change in strength from pre to post | from baseline to 8 weeks
  As many reps as possible of squats wearing a weighted vest with 20% of their bodyweight
Change in endurance from pre to post | from baseline to 8 weeks
  As long as possible in as low as possible wall sit (matching pre and post joint angles for participant)
Change in one legged strength from pre to post | from baseline to 8 weeks
  As many reps as possible standing up from a seated position on one leg and sitting back down

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Prevention Research Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided